CLINICAL TRIAL: NCT05543031
Title: Effect Of Music Integrated Phonological Awareness Program On Preschool Cochlear Implant Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Büşra Yılanlı, Research Assistant, Uskudar University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 138955
Record Dates: First submitted 2022-08-26; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Telerehabilitation
Keywords: Phonological awareness training; music; cochlear implant; telerehabilitation; mismatch negativity

STUDY DESIGN:
Intervention Model Description: This study was designed to determine the benefit of music integrated phonological awareness programs for children using cochlear implants. In addition, the phonological skills and language skills of children using cochlear implants and children with normal hearing were compared in the pre and post-training results.
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): There are 9 (35,8%) female and 14 (64,2%) male preschool cochlear implant users in the study group.
  Children ranging in age from 5 to 7 who also have 5-6 years old language skills.
  Interventions: Other: Music-Integrated Phonological Awareness training program; Diagnostic Test: Spectral-Temporally Modulated Ripple Test (SMRT); Diagnostic Test: The Phonological Awareness Scale of Early Childhood Period (PASECP); Diagnostic Test: Mismatch Negativity Test; Diagnostic Test: Early Language Development (TELD-3)
- Control group (Experimental): There are 9 (35.8%) female and 14 (64,2%) male preschool children with normal hearing in the control group.
  Children ranging in age from 5 to 6 who also have age-appropriate language skills.
  Interventions: Diagnostic Test: The Phonological Awareness Scale of Early Childhood Period (PASECP); Diagnostic Test: Early Language Development (TELD-3)

INTERVENTIONS:
Other: Music-Integrated Phonological Awareness training program — We would like to observe the effect of the music integrated phonological awareness program on preschool cochlear implant users and to compare the phonological awareness skills of the study group with the control group before and after the online training. The program is prepared as 10 lessons. Participants were guided through online training for 5 weeks, with 20-minute sessions conducted weekly. The training was carried out via Zoom, a free virtual interview program. Each family had a computer.
  Arms: Study group
Diagnostic Test: Spectral-Temporally Modulated Ripple Test (SMRT) — Spectral-Temporally Modulated Ripple Test (SMRT) was used to assess the spectral discrimination ability of the study group.Speech stimuli were presented at a calibrated presentation level of 60 dB SPL in a quiet room. The child was positioned at 0° azimuth and 1-meter from the loudspeaker.
  Arms: Study group
Diagnostic Test: The Phonological Awareness Scale of Early Childhood Period (PASECP) — The Phonological Awareness Scale of Early Childhood Period (PASECP) was used to measure the sound awareness and sound discrimination skills of study group pre-post training. The test has 8 sub-dimensions.
Diagnostic Test: Mismatch Negativity Test — Mismatch Negativity (MMN) was used to evaluate the central auditory system.The test was used for electrophysiological recordings of the study group.The standard stimulus presented as /ba/ (%80), and the rare stimulus presented as /da/ (%20) frequency. The onset (rise) and offset (fall) times of the stimuli are 10 ms, and the plateau time is 50 ms. The interval between stimuli for both responses was 1.1 ms. A 0.1-30 Hz filter was applied. The speech stimuli intensity was 70 dB SPL. Speech stimuli were presented at a 1-meter distance from the participant, with speakers placed at an angle of 0°.
  Arms: Study group
Diagnostic Test: Early Language Development (TELD-3) — Test of Early Language Development (TELD-3) measured children's receptive and expressive language skills both group for inclusion criteria.

SUMMARY:
The aim was to observe the effect of the music integrated phonological awareness program on preschool cochlear implant users and to compare the phonological awareness skills of the study group with the control group before and after the online training.

DETAILED DESCRIPTION:
This study was designed to determine the benefit of music integrated phonological awareness programs for children using cochlear implants. In addition, the phonological skills and language skills of children using cochlear implants and children with normal hearing were compared in the pre and post-training results. Test of Early Language Development (TELD-3), The Phonological Awareness Scale of Early Childhood Period (PASECP), Mismatch Negativity (MMN) was used in this study.

This study was carried out with follow-up patients in the Audiology, Language and Speech Disorders Clinic of xxx University - Medical Faculty, Department of Otorhinolaryngology. The study was performed with the approval of Ethics Committee, and written informed consent was obtained from all patient families (138955/ July 2021). There are 9 female and 14 male cochlear implant users in the study group; 9 female and 14 male children with normal hearing in the control group. Children ranging in age from 5 to 7 who also have 5-6 years old language skills without any neurological problems were included in the study. Cochlear implant mappings of all children were checked before the training.

SPSS 25.0 (IBM) was used for statistical analysis. Pre and post-training comparisons of The Phonological Awareness Scale of Early Childhood Period, SMRT, and Mismatch Negativity tests were analyzed with the Wilcoxon test. The correlation of numerical measurements with each other was examined with Spearman Correlation. The differences in the numerical measurements used in the research according to the binary demographic categories were analyzed with the Mann-Whitney U test. The differences according to the multiple categories were analyzed using the Kruskal Wallis H test. The significance level (α=0,05) was used.

ELIGIBILITY:
Inclusion Criteria:

* For children with hearing loss
* Bilateral severe sensorineural hearing loss
* Having unilateral or bilateral cochlear implants,
* Having a chronological age in the range of 5-7 years,
* Not having started primary school.
* Using the cochlear implant and regularly
* To receive regular training in the auditory rehabilitation center

For children with normal hearing:

* To have normal hearing,
* To have receptive and expressive language skills compatible with the chronological age in the language test to be performed.
* Not starting primary school

Exclusion Criteria:

* In case of not having any without being accepted for control and study,
* Having additional disability
* Using drugs affecting the auditory system

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the phonological awareness skills at 3 Months | baseline and 3 months
  The Early Childhood Phonological Awareness Scale (PASECP) was used to measure sound awareness and sound discrimination skills of preschool children whose language age is between 60-72 months. The test has 8 sub-dimensions. There are 8 test items in the first sub-dimension and 10 test items in the other sub-dimensions, with a total of 78 test items. If the answers given by the children to the scale items are correct (1), if incorrect (0), they are coded into the answer key. The test is administered to children individually. The application time for each child takes approximately 15 minutes. High scores of the child indicate that his/her phonological awareness is good.
Change from Electrophysiological at 3 Months | baseline and 3 months
  Mismatch Negativity (MMN) was used to evaluate the central auditory system. Neuron-Spectrum-5 (4/EPM) (Neurosoft, Ivanoco, Russia) was used for the electrophysiological recordings of the study group. Speech stimuli were used as stimuli. Amplitude and latency changes were observed in the Mismatch Negativity test before and after the training. The increase in amplitudes and shortening of latencies after training indicate that the central auditory system has developed.
Change from baseline in the spectral discrimination ability at 3 Months | baseline and 3 months
  Spectral-Temporally Modulated Ripple Test (SMRT) was used to assess the spectral discrimination ability of the study group. The test was performed using SMRT software. Waveform broadband noise with spectral-temporal modulation was used. In each trial, three ripple sounds were presented. Two stimuli were reference signals with an intensity of 20 ripple/octave (rpo) and another stimulus was a target signal with a lower rpo intensity. The initial intensity of the target signal was 0.5 rpo and was replaced by a step size of 0.2 rpo. Adaptive running terminated after ten reverses.Spectral-Temporally Modulated Ripple Test was calculated over the last six reversals. Three runs were completed for each child, and the final threshold was determined by averaging the three runs. Having a low rpo value was an indication of good spectral resolution of the children.

CONTACTS AND LOCATIONS:
Overall Officials: Büşra Yılanlı, Msc, Principal Investigator — Uskudar University
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul University-Cerrahpasa, Istanbul
  - Uskudar University, Istanbul

IPD SHARING:
Plan to Share IPD: No
The IPD available upon reasonable request to the other authors

REFERENCES:
- [Background] Carroll JM, Snowling MJ, Hulme C, Stevenson J. The development of phonological awareness in preschool children. Dev Psychol. 2003 Sep;39(5):913-23. doi: 10.1037/0012-1649.39.5.913. PMID 12952403
- [Background] Ching TY, Cupples L. Phonological Awareness at 5 years of age in Children who use Hearing Aids or Cochlear Implants. Perspect Hear Hear Disord Child. 2015 Sep;25(2):48-59. doi: 10.1044/hhdc25.2.48. PMID 26929789
- [Background] Ching TY, Dillon H, Katsch R, Byrne D. Maximizing effective audibility in hearing aid fitting. Ear Hear. 2001 Jun;22(3):212-24. doi: 10.1097/00003446-200106000-00005. PMID 11409857
- [Background] Soleymani Z, Mahmoodabadi N, Nouri MM. Language skills and phonological awareness in children with cochlear implants and normal hearing. Int J Pediatr Otorhinolaryngol. 2016 Apr;83:16-21. doi: 10.1016/j.ijporl.2016.01.013. Epub 2016 Jan 25. PMID 26968046
- [Result] Christiner M, Reiterer SM. Early Influence of Musical Abilities and Working Memory on Speech Imitation Abilities: Study with Pre-School Children. Brain Sci. 2018 Sep 1;8(9):169. doi: 10.3390/brainsci8090169. PMID 30200479
- [Result] Anvari SH, Trainor LJ, Woodside J, Levy BA. Relations among musical skills, phonological processing, and early reading ability in preschool children. J Exp Child Psychol. 2002 Oct;83(2):111-30. doi: 10.1016/s0022-0965(02)00124-8. PMID 12408958
- [Result] Choi JE, Won JH, Kim CH, Cho YS, Hong SH, Moon IJ. Relationship between spectrotemporal modulation detection and music perception in normal-hearing, hearing-impaired, and cochlear implant listeners. Sci Rep. 2018 Jan 15;8(1):800. doi: 10.1038/s41598-017-17350-w. PMID 29335454
- [Result] Engstrom E, Kallioinen P, Nakeva von Mentzer C, Lindgren M, Sahlen B, Lyxell B, Ors M, Uhlen I. Auditory event-related potentials and mismatch negativity in children with hearing loss using hearing aids or cochlear implants - A three-year follow-up study. Int J Pediatr Otorhinolaryngol. 2021 Jan;140:110519. doi: 10.1016/j.ijporl.2020.110519. Epub 2020 Nov 24. PMID 33268013
- [Result] DiNino M, Arenberg JG. Age-Related Performance on Vowel Identification and the Spectral-temporally Modulated Ripple Test in Children With Normal Hearing and With Cochlear Implants. Trends Hear. 2018 Jan-Dec;22:2331216518770959. doi: 10.1177/2331216518770959. PMID 29708065
- [Result] Fernandes NM, Gil D, Azevedo MF. Mismatch Negativity in Children with Cochlear Implant. Int Arch Otorhinolaryngol. 2019 Jul;23(3):e292-e298. doi: 10.1055/s-0039-1688967. Epub 2019 May 28. PMID 31360248
- [Result] Ferreira DA, Bueno CD, de Costa SS, Sleifer P. Mismatch Negativity in Children: Reference Values. Int Arch Otorhinolaryngol. 2019 Apr;23(2):142-146. doi: 10.1055/s-0038-1667313. Epub 2018 Oct 24. PMID 30956696
- [Result] Gifford RH, Noble JH, Camarata SM, Sunderhaus LW, Dwyer RT, Dawant BM, Dietrich MS, Labadie RF. The Relationship Between Spectral Modulation Detection and Speech Recognition: Adult Versus Pediatric Cochlear Implant Recipients. Trends Hear. 2018 Jan-Dec;22:2331216518771176. doi: 10.1177/2331216518771176. PMID 29716437
- [Result] Jeddi Z, Lotfi Y, Moossavi A, Bakhshi E, Hashemi SB. Correlation between Auditory Spectral Resolution and Speech Perception in Children with Cochlear Implants. Iran J Med Sci. 2019 Sep;44(5):382-389. doi: 10.30476/IJMS.2019.44967. PMID 31582862
- [Result] Jing L, Vermeire K, Mangino A, Reuterskiold C. Rhyme Awareness in Children With Normal Hearing and Children With Cochlear Implants: An Exploratory Study. Front Psychol. 2019 Sep 12;10:2072. doi: 10.3389/fpsyg.2019.02072. eCollection 2019. PMID 31572265
- [Result] Kraus N, Hornickel J, Strait DL, Slater J, Thompson E. Engagement in community music classes sparks neuroplasticity and language development in children from disadvantaged backgrounds. Front Psychol. 2014 Dec 16;5:1403. doi: 10.3389/fpsyg.2014.01403. eCollection 2014. PMID 25566109
- [Result] Landsberger DM, Padilla M, Martinez AS, Eisenberg LS. Spectral-Temporal Modulated Ripple Discrimination by Children With Cochlear Implants. Ear Hear. 2018 Jan/Feb;39(1):60-68. doi: 10.1097/AUD.0000000000000463. PMID 28682810
- [Result] Lee SAS, Hall B, Sancibrian S. Feasibility of a Supplemental Phonological Awareness Intervention via Telepractice for Children with Hearing Loss: A Preliminary Study. Int J Telerehabil. 2017 Jun 29;9(1):23-38. doi: 10.5195/ijt.2017.6216. eCollection 2017 Spring. PMID 28814992
- [Result] Linnavalli T, Putkinen V, Huotilainen M, Tervaniemi M. Phoneme processing skills are reflected in children's MMN responses. Neuropsychologia. 2017 Jul 1;101:76-84. doi: 10.1016/j.neuropsychologia.2017.05.013. Epub 2017 May 12. PMID 28506807
- [Result] Linnavalli T, Putkinen V, Lipsanen J, Huotilainen M, Tervaniemi M. Music playschool enhances children's linguistic skills. Sci Rep. 2018 Jun 8;8(1):8767. doi: 10.1038/s41598-018-27126-5. PMID 29884891
- [Result] Naatanen R, Petersen B, Torppa R, Lonka E, Vuust P. The MMN as a viable and objective marker of auditory development in CI users. Hear Res. 2017 Sep;353:57-75. doi: 10.1016/j.heares.2017.07.007. Epub 2017 Jul 20. PMID 28800468
- [Result] Ni G, Zheng Q, Liu Y, Zhao Y, Yue T, Han S, Liu H, Ming D. Objective electroencephalography-based assessment for auditory rehabilitation of pediatric cochlear implant users. Hear Res. 2021 May;404:108211. doi: 10.1016/j.heares.2021.108211. Epub 2021 Feb 18. PMID 33684887
- [Result] Patscheke H, Dege F, Schwarzer G. The Effects of Training in Music and Phonological Skills on Phonological Awareness in 4- to 6-Year-Old Children of Immigrant Families. Front Psychol. 2016 Oct 21;7:1647. doi: 10.3389/fpsyg.2016.01647. eCollection 2016. PMID 27818643
- [Result] Scott JA, Goldberg H, Connor CM, Lederberg AR. Schooling Effects on Early Literacy Skills of Young Deaf and Hard of Hearing Children. Am Ann Deaf. 2019;163(5):596-618. doi: 10.1353/aad.2019.0005. PMID 30713200
- [Result] Soleimanifar S, Jafari Z, Motasaddi Zarandy M, Asadi H, Haghani H. Relationship between Intelligence Quotient and Musical Ability in Children with Cochlear Implantation. Iran J Otorhinolaryngol. 2016 Sep;28(88):345-352. PMID 27738611
- [Result] Torppa R, Faulkner A, Laasonen M, Lipsanen J, Sammler D. Links of Prosodic Stress Perception and Musical Activities to Language Skills of Children With Cochlear Implants and Normal Hearing. Ear Hear. 2020 Mar/Apr;41(2):395-410. doi: 10.1097/AUD.0000000000000763. PMID 31397704
- [Result] Wang Y, Liu L, Zhang Y, Wei C, Xin T, He Q, Hou X, Liu Y. The Neural Processing of Vocal Emotion After Hearing Reconstruction in Prelingual Deaf Children: A Functional Near-Infrared Spectroscopy Brain Imaging Study. Front Neurosci. 2021 Jul 28;15:705741. doi: 10.3389/fnins.2021.705741. eCollection 2021. PMID 34393716
- [Result] Webb MY, Lederberg AR. Measuring phonological awareness in deaf and hard-of-hearing children. J Speech Lang Hear Res. 2014 Feb;57(1):131-42. doi: 10.1044/1092-4388(2013/12-0106). PMID 23900033
- [Result] Won JH, Clinard CG, Kwon S, Dasika VK, Nie K, Drennan WR, Tremblay KL, Rubinstein JT. Relationship between behavioral and physiological spectral-ripple discrimination. J Assoc Res Otolaryngol. 2011 Jun;12(3):375-93. doi: 10.1007/s10162-011-0257-4. Epub 2011 Jan 27. PMID 21271274
- See also: Davis, M. M. (2019). Rhythms and Reading : Applying Literacy to the Music Classroom. — http://encompass.eku.edu/honors_theses/613
- See also: DuBois, G. E. (2021). Using Group Music Activities with Families to Support School-Readiness Skills in Preschool Children with Hearing Loss. ProQuest Dissertations and Theses, 6(1), 160. — http://www.proquest.com/dissertations-theses/using-group-music-activities-with-families/docview/2556426431/se-2?accountid=135034
- See also: Phelps, S. (2003). Phonological Awareness Training in a Preschool Classroom of Typically Developing Children. Electronic Theses and Dissertations. — http://dc.etsu.edu/etd/772
- See also: Eissa, M. A. (2013). The Effectiveness of a Phonological Awareness Training Intervention on Pre-reading Skills of Children with Mental Retardation. Psycho-Educational Research Reviews, 2(2), 11-21. — http://perrjournal.com/index.php/perrjournal/article/view/377
- Available data/document: Study Protocol — http://dc.etsu.edu/etd/772
- Available data/document: Study Protocol — http://encompass.eku.edu/honors_theses

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT05543031/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT05543031/ICF_001.pdf